CLINICAL TRIAL: NCT01411709
Title: A Pilot Study On The Effect Of Vitano® On Physiological And Psychological Responses To Psychological Stress Assessed Under Laboratory Conditions And In Everyday Life
Brief Title: A Study On The Effect Of Vitano® On Physiological And Psychological Responses To Psychological Stress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Dr. Willmar Schwabe GmbH & Co. KG (Industry)
Responsible Party: Dr Hubert Bland, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC287
Record Dates: First submitted 2011-07-28; First posted 2011-08-08 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Mild Stress/Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitano (Active Comparator)
  Interventions: Drug: Vitano
- Control (No Intervention): No tablets - control group

INTERVENTIONS:
Drug: Vitano — two 200mg tablets per day for 14 days
  Arms: Vitano

SUMMARY:
A pilot investigation into the stress relieving properties of Vitano® which will assess the following hypotheses

Individuals exposed to Vitano® will demonstrate diminished blood pressure and heart rate responses to mental stress compared to individuals in the control condition

Physiological recovery (BP, HR and cortisol) from mental stress will be enhanced in individuals exposed to Vitano® compared to individuals in the control condition

Vitano® will have positive effects on cognitive functioning.

Subjective ratings of stress will be reduced in individuals exposed to Vitano® compared to individuals in the control condition

There will be a significant improvement in subjective well-being in individuals taking Vitano®.

ELIGIBILITY:
Inclusion Criteria:

* subject is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
* The subject has signed the ICF.
* Healthy male or female subjects aged 18-35 years inclusive. Attempts will be made to achieve an equal gender ratio through appropriate screening procedures, but a failure to do so will not preclude analysis of the final data set.
* A score above 30 on the Spielberger State-Trait Anxiety Inventory (STAI).
* The subject agrees to use suitable methods of contraception during the study and for 3 months afterwards.
* The subject is a non-smoker.
* The subject is, in the opinion of the Investigator, healthy on the basis of medical history, vital signs, and the results of routine laboratory tests.

Exclusion Criteria:

* The subject is pregnant or breast feeding.
* The subject consumes more than 5 caffeine-containing beverages per day.
* The subject is colour blind.
* Clinically significant hepatic or renal abnormality as determined by laboratory tests.
* BMI above 33.
* History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1.
* Positive alcohol breath test at any visit. A repeat test will not be allowed. [NOTE: subjects must be told to avoid consumption of alcoholic beverages for at least 24 hours prior to attending the Centre].
* Use of any other medication which may interfere with study outcome and/or interfere with IMP within the 2 weeks or 5 half lives preceding the first treatment phase, with the exception of contraceptive pill, non-steroidal analgesics, and paracetamol. [NOTE: Concomitant medications which do not influence study outcome and/or do not interfere with IMP may be allowed at the discretion of the Investigator].
* Current participation in another clinical trial with an investigational or non-investigational drug or device, or participation in another clinical trial within the 3 months preceding Visit 1 (screening visit).
* Any condition that, in the Investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
* Moderate or severe anxiety* *If participants are found to have moderate or severe anxiety during the screening process then they will be referred to the University Counselling service.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurements | Measurements over 14 days (Day 0, Day 7 and Day 14)
  Blood pressure readings taken under laboratory conditions during cognitive testing and relaxation periods

SECONDARY OUTCOMES:
Measures of cognitive function | 14 days
  cognitive function assessed four times during the 14 day study period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom